CLINICAL TRIAL: NCT01386619
Title: Natural Killer Cell Selected T-cell Depleted Donor Lymphocyte Infusions (NK-DLI) in Patients After HLA-haploidentical Allogeneic Stem Cell Transplantation
Brief Title: NK DLI in Patients After Human Leukocyte Antigen (HLA)-Haploidentical Hematopoietic Stem Cell Transplantation (HSCT)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK-DLI Allo-Tx
Record Dates: First submitted 2011-06-07; First posted 2011-07-01 (Estimated); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Lymphoma; Neuroblastoma; Rhabdomyosarcoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Lymphoma; Neuroblastoma; Rhabdomyosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NK cell DLI (Experimental)
  Interventions: Biological: CD3-depleted/CD56+ selected natural killer cells collected from apheresis products

INTERVENTIONS:
Biological: CD3-depleted/CD56+ selected natural killer cells collected from apheresis products — NK DLI products containing >1 10e7 NK cells/kg bodyweight (BW) and < 1 x 10e5 T-cells/kg BW are administered at days +4 (Frankfurt only), and on days +40 and +100 (both centers)

SUMMARY:
This is a phase I/II study of highly selected donor lymphocyte infusions in patients undergoing HLA-haploidentical hemopoietic stem cell transplantation. Patients will be offered "pre-emptive" NK-DLI early after HSCT.

Three schedules of NK-cell infusion will be studied: Basel patients (adult and pediatric) will receive NK-DLI on days +40 and +100 (pre-emptive-late); Frankfurt patients (pediatric) will receive NK-DLI on days +3, +40, and +100 (pre-emptive early). Patients not receiving pre-emptive NK-DLI with loss in donor chimerism or with evidence of minimal residual disease will be offered "therapeutic" NK-DLI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute/chronic leukemia, myelodysplastic syndrome, lymphoid neoplasia, solid tumor or bone marrow failure syndrome
* signed informed consent of the patient (or his/her legal representative)

Exclusion Criteria:

* Patients with graft failure
* Patients with any grade of active acute of chronic graft-versus-host disease (GvHD)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Feasibility of NK-DLI production | At day of transplant (day 0)
  The feasibility of the production of expanded NK-cell DLI will be measured. Primary quality measures of the NK cell product are the number of NK cells that can be produced (CD56+/cluster of differentiation 3(CD3)- NK cell goal dose >= 1 * 10e7/kg body weight of recipient) as well as the degree of CD3 T-cell contamination (goal CD3+ T-cell dose < 1 * 10e5 / kg body weight of recipient).
Safety of NK DLI Infusion | Day +60 after transplant
  The safety evaluation regards transfusion associated adverse events (fever, fall in blood pressure, transfusion site reactions, etc) and is evaluated at the time of NK DLI infusion. The primary long-term safety measure is the absence of acute graft-versus-host disease 30 days after the last NK DLI infusion.

SECONDARY OUTCOMES:
Efficacy of NK DLI Infusions | 5 years after last NK DLI
  The efficacy of NK DLI infusions will be assessed by evaluation of the rates of overall and disease free survival and the rate of disease relapse. As this is a single arm study, outcome measures assessed will be compared to those of historical controls treated with haploidentical HSCT without NK DLI infusions.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Passweg, MD, Study Chair — University Hospital, Basel, Switzerland; Dirk Schwabe, MD, Study Chair — Johann Wolfgang Goethe University Hospital
Locations (2):
- Universitätsklinikum, Frankfurt, Germany
- University Hospital, Basel, Switzerland